CLINICAL TRIAL: NCT01006681
Title: Efficacy and Safety of Vaccination Against Influenza H1N1 in Patients With Rheumatoid Arthritis, Systemic Lupus Erythematosus, Psoriatic Arthritis and Ankylosing Spondylitis Treated With Immunomodulatory Drugs
Brief Title: Vaccination Against Influenza H1N1 in Rheumatic Diseases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Ori Elkayam, Tel Aviv Sourasky Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0560-09
Record Dates: First submitted 2009-10-31; First posted 2009-11-03 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Influenza; Rheumatic Diseases
Keywords: rheumatoid; SLE; Psoriatic arthritis; Ankylosing; Influenza H1N1; Vaccine; Vaccination against H1N1 in rheumatic diseases
MeSH Terms: conditions — Influenza, Human; Rheumatic Diseases; Arthritis, Psoriatic | interventions — focetria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Monovalent MF59-Adjuvanted vaccine (Experimental)
  Interventions: Biological: Focetria (Monovalent MF59-Adjuvanted vaccine)

INTERVENTIONS:
Biological: Focetria (Monovalent MF59-Adjuvanted vaccine) — 7.5 mcg Hemagglutinin H1/InfluezaA/California/7/2009 ,9.75 mg squalene MF59, 1.175 mg polysort80, 1.175 mg sorbitan trioleate
  Intra muscular
  Other Names: Focetria
Biological: Focetria (Monovalent MF59-Adjuvanted vaccine) — 7.5 mg Hemagglutinin H1/InfluezaA/California/7/2009, 9.75 mg squalene MF59, 1.175 mg polysirate 80, 1.175 mg sorbitan trioleate
  Intramuscular injection
  Other Names: Focetria
Biological: Focetria (Monovalent MF59-Adjuvanted vaccine) — Monovalent MF59-Adjuvanted vaccine
  Other Names: Focetria

SUMMARY:
The spread of Influenza H1N1 has prompted the development of vaccines against this virus. Immunocompromised patients are at increased risk of developing complications of Influenza H1N1. The efficacy and safety of H1N1 vaccination have not been evaluated in this population of patients.

DETAILED DESCRIPTION:
100 patients with Rheumatoid Arthritis (RA), 50 patients with Systemic Lupus Erythematosus (SLE), 50 patients with spondyloarthropathies (Psoriatic arthritis (PsA) and Ankylosing Spondylitis (AS) and 200 healthy subjects will participate in the study.

All the subjects will be vaccinated with Focetria (Novartis) and will be evaluated the day of vaccination and 4 weeks later.

The evaluation will include:

Efficacy of the vaccine: Blood will be drawn on day 0 and 4 weeks later and tested for the presence of antibodies against A/California17/2009/H1N1 by hemagglutination inhibition test.

Safety of the vaccine:

* Records of adverse event
* Assessment of disease activity : RA - Disease activity score (DAS 28), SLE - SLEDAI, PsA - DAS 28 and PASI, AS- BASDAI, ESR, CRP

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from: Rheumatoid Arthritis, Systemic Lupus Erythematosus, Ankylosing Spondylitis, Psoriatic Arthritis
* Able to firm an informed consent
* Aged - 18-65
* Candidates to receive vaccination against H1N1, according to the recommendation of the Ministry of Health

Exclusion Criteria:

* Allergy to eggs
* Known allergy to seasonal influenza vaccine
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-04 (Estimated); Study Completion 2010-04 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint : Proportion of patients who will achieve a titer of antibodies above 1/40 within the groups of patients in comparison with healthy subjects | 4 weeks

SECONDARY OUTCOMES:
Secondary Endpoint: Safety of the vaccine with regard to disease activity by changes in DAS, SLEDAI and BASDAI | 4 weeks

REFERENCES:
- [Derived] Elkayam O, Amir S, Mendelson E, Schwaber M, Grotto I, Wollman J, Arad U, Brill A, Paran D, Levartovsky D, Wigler I, Caspi D, Mandelboim M. Efficacy and safety of vaccination against pandemic 2009 influenza A (H1N1) virus among patients with rheumatic diseases. Arthritis Care Res (Hoboken). 2011 Jul;63(7):1062-7. doi: 10.1002/acr.20465. PMID 21425247